CLINICAL TRIAL: NCT07211022
Title: Clinical Evaluation of the Complete Arch Digital Impressions Accuracy Using Photogrammetry and Intraoral Scanning
Brief Title: Precision of Digital Impressions in Complete-Arch Implant Rehabilitation: Evaluation of Two Digital Techniques
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aldent University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DIGIMP-FULLARCH-2025-01
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Complete Edentulism
Keywords: digital impression; photogrammetry; Intraoral scanning

STUDY DESIGN:
Intervention Model Description: This is a cross over in vivo clinical study in which each participant will undergo both digital impressions IOS and Intraoral Photogrammetry , using conventional impression technique as reference.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intraoral Scanner (Active Comparator): Digital scanning of edentulous arches using intraoral scanner (Aoralscan Elite, Shining 3D)
  Interventions: Procedure: Digital impression using intraoral scanner
- Intraoral Photogrammetry (Active Comparator): Digital scanning of edentulous arches using intraoral photogrammetry (Aoralscan Elite, Shining 3D)
  Interventions: Procedure: Digital impression using intraoral photogrammetry
- Conventional impression of edentulous arches (Active Comparator): Conventional impression of complete- arch edentulous patients
  Interventions: Procedure: Conventional impression

INTERVENTIONS:
Procedure: Digital impression using intraoral scanner — Digital impression of complete- arch edentulous patients using intraoral scanner
  Arms: Intraoral Scanner
Procedure: Digital impression using intraoral photogrammetry — Digital impression of complete-arch edentulous patients using intraoral photogrammetry
  Arms: Intraoral Photogrammetry
Procedure: Conventional impression — Conventional impression of complete-arch edentulous patients
  Arms: Conventional impression of edentulous arches

SUMMARY:
This clinical trial evaluates the accuracy of two digital impression techniques intraoral photogrammetry and intraoral scanning in patients rehabilitated with full-arch implant-supported prostheses (All-on-4 and All-on-6 concepts).

DETAILED DESCRIPTION:
The study aims to evaluate and compare two digital impression techniques, intraoral scanning and intraoral photogrammetry methods in terms of precision, accuracy (using conventional impression technique as reference), and virtual fit of complete-arch implant supported restorations. The trial is an in vivo cross over study with direct 3D deviation analysis and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* Edentulous maxilla or mandible
* All-on-4 or All-on-6 implant supported restoration
* Ability to provide informed consent

Exclusion Criteria:

* Severe systemic diseases (ASA III+)
* Bisphosphonate therapy
* Heavy bruxism
* Inability to attend follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-01-25 (Actual); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Digital impressions of all the enrolled patients | After 3 months from implant placement for all the enrolled patients
  STL files of digital impressions, intraoral scanning and photogrammetry , of all the enrolled patients.

SECONDARY OUTCOMES:
Virtual analyses of implant positions | Within 3 months from digital impression
  3D deviation between implant positions captured by intraoral scanning vs. intraoral photogrammetry digital impression - measured using metrology software (Geomagic Control X)

CONTACTS AND LOCATIONS:
Overall Officials: Brunilda Koci, Assoc. Prof., Principal Investigator — Aldent University
Locations (1):
- University Dental Clinic of Aldent University, Tirana, Albania, Albania

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol
Time Frame: The full study protocol will be made available beginning 1 year after publication of the primary results in a peer-reviewed journal and ending 2 years after the publication of results.
Access Criteria: The full study protocol will be shared upon reasonable request to qualified researchers . Requests should be submitted to the principal investigator via institutional email. Data will be provided after approval of the proposal and completion of a data agreement to ensure appropriate use of the data. Shared files will be transmitted through a secure institutional repository.

REFERENCES:
- See also: Precision of complete-arch digital implant scans using photogrammetry and intra-oral scanning. An in vivo cross-over study — https://pubmed.ncbi.nlm.nih.gov/40545227/